CLINICAL TRIAL: NCT01576653
Title: Prospective Clinical Evaluation of Bata-D-Glucan Assay for Diagnosis of Invasive Fungal Infection in Blood and Bronchoalveolar Lavage
Brief Title: Prospective Clinical Evaluation of Beta-D-Glucan Assay in Blood and BAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Krause, MD (Other)
Responsible Party: Sponsor-Investigator, Robert Krause, MD, MD, Medical University of Graz
Organization: Medical University of Graz (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-343
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Invasive Fungal Infection; Hematological Malignancy; Receipt of Solid Organ Transplant
Keywords: IFI
MeSH Terms: conditions — Invasive Fungal Infections; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No IFI (Active Comparator): Bronchoscopy will be performed routinely in most patients with clinical suspicion of IFI. IFIs in patients will be retrospectively graded in possible, probable, proven and no IFI according to revised EORTC/MSG criteria. Patients that do not fulfill EORTC/MSG IFI criteria will serve as negative controls.
  Interventions: Other: Fungitell Assay in BAL
- IFI (Active Comparator): Bronchoscopy will be performed routinely in most patients with clinical suspicion of IFI. IFIs in patients will be retrospectively graded in possible, probable, proven and no IFI according to revised EORTC/MSG criteria. Patients that do fulfill EORTC/MSG criteria of possible/probable/proven IFI will serve as study group.
  Interventions: Other: Fungitell Assay in BAL

INTERVENTIONS:
Other: Fungitell Assay in BAL — Fungitell Assay will be performed in BAL from patients with clinical suspicion of IFI

SUMMARY:
In patients with invasive fungal infection (IFI) rapid diagnosis is essential for early initiation of appropriate antifungal therapy and thereby survival. Conventional culture is still the Gold-Standard for diagnosis of IFI. Sensitivity of conventional culture, however, is low (50%) and time to results minimum 24 hours.

Therefore usage of serological tests detecting fungal antigens has increased dramatically over recent years. Main advantages of this new methods are rapid results and higher sensitivity when compared to conventional culture. One of the most promising serological marker currently used is beta-D-Glucan, which is a component of the fungal cell wall. ß-D-Glucan has been detected in IFI caused by Aspergillus, Candida and Fusarium spp. The Fungitell Assay (Associates of Cape Code, Inc.) was developed and validated for detection of ß-D-Glucan in peripheral blood.

Up to date information about clinical performance of the Fungitell Assays in bronchoalveolar lavage fluid (BAL) is limited. This study will therefore evaluate clinical and diagnostic performance of the Fungitell Assay in BAL from patients with solid organ transplant or hematologic malignancy.

In addition Mn/A-Mn, the lateral flow device test for aspergillosis, and Galactomannan, as well as PCR will be determined and used as comparators for BDG performance.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* Bronchoscopy performed in clinical routine due to suspicion of IFI
* Hematological malignancy or receipt of solid organ transplant/ICU

Exclusion Criteria:

* below 18 years of age
* No bronchoscopy performed
* No Hematological malignancy nor receipt of solid organ transplant/ICU

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Fungitell Assay from BAL in patients with hematologic malignancy or ICU patients/patients after solid organ transplantation and suspected IFI | 6 months after intervention
  Diagnostic potential of Fungitell Assay from BAL in patients with hematologic malignancy or ICU patients/ patients after solid organ transplantation and suspected IFI

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Prattes J, Raggam RB, Vanstraelen K, Rabensteiner J, Hoegenauer C, Krause R, Pruller F, Wolfler A, Spriet I, Hoenigl M. Chemotherapy-Induced Intestinal Mucosal Barrier Damage: a Cause of Falsely Elevated Serum 1,3-Beta-d-Glucan Levels? J Clin Microbiol. 2016 Mar;54(3):798-801. doi: 10.1128/JCM.02972-15. Epub 2015 Dec 30. PMID 26719433
- [Derived] Reischies FM, Raggam RB, Prattes J, Krause R, Eigl S, List A, Quehenberger F, Strenger V, Wolfler A, Hoenigl M. Urine Galactomannan-to-Creatinine Ratio for Detection of Invasive Aspergillosis in Patients with Hematological Malignancies. J Clin Microbiol. 2016 Mar;54(3):771-4. doi: 10.1128/JCM.02969-15. Epub 2015 Dec 23. PMID 26699701
- [Derived] Prattes J, Hoenigl M, Rabensteiner J, Raggam RB, Prueller F, Zollner-Schwetz I, Valentin T, Honigl K, Fruhwald S, Krause R. Serum 1,3-beta-d-glucan for antifungal treatment stratification at the intensive care unit and the influence of surgery. Mycoses. 2014 Nov;57(11):679-86. doi: 10.1111/myc.12221. Epub 2014 Jul 15. PMID 25040144